CLINICAL TRIAL: NCT02813486
Title: Safety and Immunogenicity Study of Tetanus, Diphtheria and Acellular Pertussis (Tdap) Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3111_P1/2a
Record Dates: First submitted 2016-06-20; First posted 2016-06-27 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Tetanus; Diphtheria; Whooping Cough
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GC3111 Vaccine Group (Experimental): Participants randomized to receive a single dose of GC3111 vaccine (Biological: GC3111 vaccine).
  Interventions: Biological: Biological: GC3111 vaccine
- Boostrix® Vaccine Group (Active Comparator): Participants randomized to receive a single dose of Boostrix® vaccine (Biological: Boostrix® vaccine).
  Interventions: Biological: Biological: Boostrix® vaccine

INTERVENTIONS:
Biological: Biological: GC3111 vaccine — 0.5mL, Intramuscular
  Other Names: GC3111
  Arms: GC3111 Vaccine Group
Biological: Biological: Boostrix® vaccine — 0.5mL, Intramuscular
  Other Names: Boostrix®
  Arms: Boostrix® Vaccine Group

SUMMARY:
The purpose of this study is to evaluate safety of GC3111 and to describe immunogenicity of a single dose of GC3111 versus Boostrix® vaccine among healthy adults in 19 to <65 years of age.

DETAILED DESCRIPTION:
To evaluate immunogenicity of GC3111 as tetanus, diphtheria and acellular pertussis (Tdap) vaccine in healthy adults.

To evaluate safety (solicited adverse events) of GC3111 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged between 19 and 64 years at the time of vaccination
* Informed consent and assent forms have been signed and dated

Exclusion Criteria:

* Known or suspected receipt of any Tdap vaccine
* Subject is pregnant, or lactating, or of child bearing potential without using an effective method of contraception or not practicing abstinence
* Receipt of any vaccine within 30 days before receiving study vaccine
* Any condition that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Participants With Antibody Responses to Tetanus and Diphtheria Components Following Vaccination With Either GC3111 or Boostrix® Vaccine | Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Percentage of Participants Achieving Predefined Antibody Level for Diphtheria, Tetanus, and Acellular Pertussis Antigens | 28 days after Vaccination
Geometric Mean Concentrations (GMC) for Diphtheria, Tetanus and Acellular Pertussis Antigens | 28 days after Vaccination
Geometric Mean Ratio (GMR) of post-vaccination versus pre-vaccination antibody concentrations against Diphtheria, Tetanus and Acellular Pertussis | Day 0 (pre-vaccination) to Day 28 (post-vaccination)

SECONDARY OUTCOMES:
Participants Reporting Immediate Solicited Adverse Events Following Vaccination With Either GC3111 or Boostrix® Vaccine | Up to 30 minutes post-vaccination

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Incheon St. Mary's Hospital Catholic Univ., Incheon, Bupyeong 6-dong, Bupyeong-gu,
  - The Catholic Univ. of Korea Daejeon St.Mary's Hospital, Daejeon, Jung-Gu
  - The Catholic Univ.of Korea Bucheon St.Mary's Hospital, Gyeonggi-do
  - The Catholic Univ.of Korea Uijeongbu St.Mary's Hospital, Gyeonggi-do
  - The Catholic Univ.of Korea Yeouido St.Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No